CLINICAL TRIAL: NCT01330238
Title: Phase 2 Study of the Efficacy of Zoledronic Acid in Low Back Pain Related to Vertebral Endplate Signal Changes, the So-called Modic Changes
Brief Title: The Efficacy of Zoledronic Acid in Modic Changes-related Low Back Pain (LBP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Katri Koivisto, Specialist in Physical and Rehabilitation Medicine, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT 2008-005351-14
Record Dates: First submitted 2011-02-11; First posted 2011-04-06 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Low Back Pain
Keywords: Low back pain; Modic changes; Vertebral endplate signal changes; Efficacy; Zoledronic acid; Bisphosphonates; RCT
MeSH Terms: conditions — Low Back Pain | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zoledronic acid (Active Comparator): Single infusion of 5 mg zoledronic acid I.V.
  Interventions: Drug: Zoledronic acid vs. placebo
- Placebo (Placebo Comparator): Single infusion of 100 ml isotonic NaCl-solution I.V.
  Interventions: Drug: Zoledronic acid vs. placebo

INTERVENTIONS:
Drug: Zoledronic acid vs. placebo — Single infusion of zoledronic acid or placebo
  Other Names: Aclasta; Zometa

SUMMARY:
Modic changes are associated with low back pain (LBP) both in clinical and general population-based samples. Type I changes are regarded as more likely to be painful than type II changes. Several studies suggest that type I changes are inflammatory in nature.

DETAILED DESCRIPTION:
So far, no treatment exists for LBP due to Modic changes. Bisphosphonates could be effective in this specific low back disorder through two mechanisms: 1) they could consolidate vertebral bodies thereby improving the tolerance for mechanical load and 2) they could diminish inflammation as observed recently in case of ibandronate in an experimental model.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years old
* low back pain for more than 3 months
* Modic type I or II change in lumbar magnetic resonance imaging
* Intensity of low back pain at least 6 on 10-cm VAS or Oswestry disability score at least 30%

Exclusion Criteria:

* premenopausal female patients with possibility of pregnancy
* patients with calculated creatinine clearance of less than 40 ml/min
* patients with hypocalcemia
* patients with known hypersensitivity to zoledronic acid or other bisphosphonates or ingredients of the infusional product
* patients with red flags symptoms
* patients with nerve root impingement
* patients with willingness for early retirement

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-12; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Low back pain (VAS) | 0, 1, 12 months

SECONDARY OUTCOMES:
Health-related quality of life (RAND-36) | 0, 1, 12 months
Flexibility of the lumbar spine | 0, 1, 12 months
  Modified Schober measure
Sick leaves | 0, 12 months
  Patient-reported
Radiologic phenotype | 0, 12 months
  Change in proportion and size of type I changes
Disability (Oswestry) | 0, 1, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jaro Karppinen, Prof, Study Chair — University of Oulu; Katri Koivisto, MD, Principal Investigator — University of Oulu; Eero Kyllönen, MD, Study Director — University Hospital of Oulu; Kaj Sundqvist, MD, Study Director — University Hospital of Oulu; Jaakko Niinimäki, MD, Study Director — University of Oulu; Osmo Tervonen, Prof., Study Director — University of Oulu
Locations (1):
- Institute of Clinical Sciences, Department of Physical and Rehabilitation Medicine, University of Oulu, Oulu, Finland

REFERENCES:
- [Derived] Koivisto K, Jarvinen J, Karppinen J, Haapea M, Paananen M, Kyllonen E, Tervonen O, Niinimaki J. The effect of zoledronic acid on type and volume of Modic changes among patients with low back pain. BMC Musculoskelet Disord. 2017 Jun 23;18(1):274. doi: 10.1186/s12891-017-1632-z. PMID 28645291
- [Derived] Koivisto K, Kyllonen E, Haapea M, Niinimaki J, Sundqvist K, Pehkonen T, Seitsalo S, Tervonen O, Karppinen J. Efficacy of zoledronic acid for chronic low back pain associated with Modic changes in magnetic resonance imaging. BMC Musculoskelet Disord. 2014 Mar 4;15:64. doi: 10.1186/1471-2474-15-64. PMID 24588905